CLINICAL TRIAL: NCT04976894
Title: Korean Stroke Cohort for Functioning and Rehabilitation-II
Acronym: KOSCO-II
Status: Active, not recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Yun-Hee Kim, Professor, Samsung Medical Center
Other Study IDs: 2019-11-095
Record Dates: First submitted 2021-07-16; First posted 2021-07-26 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Stroke
Keywords: Stroke; Disability; Function; Rehabilitation; Burden
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: open — open

SUMMARY:
Korean Stroke Cohort for functioning and rehabilitation (KOSCO)-II is a large, multi-centre prospective cohort study for all acute first-ever stroke patients admitted to participating hospitals in nine distinct areas of Korea. This study is designed as a 10-year, longitudinal follow-up investigating the residual disabilities, activity limitations, and quality of life issues arising in patients suffering from first-ever stroke as previous similar stroke cohort with KOSCO. The main objectives of this study are to identify and compare the factors that influence residual disability and long-term quality of life in first-ever acute stroke patients with KOSCO. The secondary objectives of this study are to determine and compare the risk of mortality and recurrent vascular events in first-ever acute stroke patients with KOSCO. Investigators will investigate longitudinal health behaviors and patterns of healthcare utilization, including stroke rehabilitation care. Investigators will also investigate the long-term health status, mood, and quality of life in stroke patient caregivers. In addition, investigators will identify baseline and ongoing characteristics that are associated with secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* First-ever acute stroke (ischemic stroke or intracerebral hemorrhage) with corresponding lesion and/or evidence of acute arterial occlusion on CT (A)- or MRI/A-scan.
* Age ≥ 19 years at onset of stroke.
* Onset of symptoms within seven days prior to inclusion.

Exclusion Criteria:

* Transient ischemic attack.
* History of stroke.
* Traumatic intracerebral hemorrhage.
* Not Korean.

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All consecutive patients with an acute first-ever stroke, admitted to the representative hospitals in the nine distinct areas of Korea, will be asked to participate in the study. Participating study centres are Samsung Medical Center, Seoul; Severance Hospital, Seoul; Konkuk University Hospital, Seoul; Chungnam National University Hospital, Daejeon; Chonnam National University Hospital, Gwangu; Pusan National University Yangsan Hospital, Yangsan; Kyungpook National University Hospital, Deagu; Wonkwang University Hospital, Iksan; and Jeju National University Hospital, Jeju.
Sampling Method: Non-Probability Sample
Enrollment: 2431 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Korean modified Barthel Index | 3 months, 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months, 72 months, 84 months, 96 months, 108 months after stroke onset.
  measurement for activities of daily living Minimum: 0, Maximum: 100 Higher scores means a better.
Change in Euro Quality of Life-5 Dimensions measurement for quality of life | 3 months, 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months, 72 months, 84 months, 96 months, 108 months after stroke onset.
  measurement for quality of life Minimum: 0, Maximum: 1 Higher scores means a better.
Change in Functional Independence Measurement | 3 months, 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months, 72 months, 84 months, 96 months, 108 months after stroke onset.
  measurement for activities of daily living Minimum: 0, Maximum: 126 Higher scores means a better.
Change in Korean Mini-Mental State Examination | 7 days, 3 months, 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months, 72 months, 84 months, 96 months, 108 months after stroke onset.
  measurement for language function Minimum: 0, Maximum: 30 Higher scores means a better.
Change in Korean Version of Frenchay Aphasia Screening Test | 7 days, 3 months, 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months, 72 months, 84 months, 96 months, 108 months after stroke onset.
  measurement for language function Minimum: 0, Maximum: 30 Higher scores means a better.
Change in modified Rankin Scale | 7 days, 3 months, 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months, 72 months, 84 months, 96 months, 108 months after stroke onset
  Measurement for disability. Range of total score 0 to 6. 0 is no disability at all and 6 is death. Therefore, greater value means worse functional status
Change in American Speech-Language-Hearing Association National Outcome Measurement System Swallowing Scale | 7 days, 3 months, 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months, 72 months, 84 months, 96 months, 108 months after stroke onset
  Measurement for swallowing function. Range of scale is 0 to 7, and greater value means better function. For example, 7 means no swallowing difficulty at all.
Change in Geriatric depression scale-short form | 3 months, 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months, 72 months, 84 months, 96 months, 108 months after stroke onset
  measurement for depression. The scale is 0 to 15. 0 is normal whereas 15 indicates severe depression.
  Minimum: 0, Maximum: 15. Lower scores means a better.
Change in Functional Ambulatory Category | 7 days, 3 months, 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months, 72 months, 84 months, 96 months, 108 months after stroke onset
  measurement for gait function Minimum: 0, Maximum: 5 Higher scores means a better.

CONTACTS AND LOCATIONS:
Overall Officials: Yun-Hee Kim, MD.,PhD., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No